CLINICAL TRIAL: NCT01116843
Title: A Preoperative Window of Opportunity Study to Assess the Modulation of Biomarkers in the Primary Tumor Site of Patients With Resectable Oral Cavity Cancer (OCC) Randomized to Receive Preoperative Treatment With PF-00299804
Brief Title: Study to Assess Biomarkers in Patients With Resectable Oral Cavity Cancer Randomized to Receive Preoperative Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WS590266
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Oral Cavity Cancer
Keywords: Oral cavity cancer; No prior treatment
MeSH Terms: conditions — Mouth Neoplasms | interventions — dacomitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF-00299804 (Experimental): Patient will receive PF-00299804 pre-operatively at a dose of 45 mg once daily orally for 7-11 days depending on surgery schedule.
  Interventions: Drug: PF-00299804
- Placebo arm (Placebo Comparator): Patient will receive matching Placebo for 7-11 days depending on surgery schedule.
  Interventions: Drug: PF-00299804

INTERVENTIONS:
Drug: PF-00299804 — PF-00299804 or Placebo given pre-operatively for 7 to 11 days depending on surgery schedule.
  Other Names: A7471001

SUMMARY:
The objective of this study is to assess the biological effects in the primary tumor following a short, pre-operative course of treatment with PF-00298804 in patients with Oral Cavity Cancer.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blinded, biomarker driven, preoperative window of opportunity study with a pharmacodynamic primary endpoint. Patients with resectable, histologically confirmed OCC for whom surgical treatment is planned as definitive management, will be randomized 2:1 to receive PF-00299804 pre-operatively at a dose of 45 mg once daily orally for 7-11 days or to Matching Placebo for 7-11 days depending on surgery schedule. The target is a total of 8 days of treatment but with a minimum of 7 and a maximum of 11 dosing days. All patients will receive surgery as per standard of care without delay. Biomarkers from the surgical specimen and baseline tumor biopsy or consent to provide a tumor block from existing primary diagnostic tumor biopsy completed within 90 days will be evaluated for primary and secondary pharmacodynamic endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Signed, voluntary informed consent provided
* Willing and able to comply with scheduled visits, treatment plan, tests, other study procedures
* Patient must be diagnosed with histologically confirmed oral cavity squamous cell carcinoma (OCC) (lip, floor of mouth, anterior 2/3 tongue, buccal mucosa, upper and lower gingiva, hard palate and retromolar trigone) considered resectable (T1-4a, N0-2, M0; (without distant metastases)) for whom surgical resection of tumor is planned. Patients with distant metastatic disease or diagnosis of SCCHN may not be enrolled
* Must be able to provide a fresh tumor biopsy prior to randomization for histopathological and biomarker evaluation. No anti-neoplastic treatment allowed between obtaining baseline tumor specimen and randomization. Patients who decline an in-house fresh pre-treatment tumor biopsy must give consent to provide a tumor block from an existing diagnostic primary tumor biopsy completed within 90 days of enrolment
* Prior treatment with agents targeted to epidermal growth factor receptor is not allowed.
* No prior chemotherapy or radiotherapy (to primary site/nodes).
* Patient must not have received prior anti-neoplastic treatment within past 2 years
* Any treatment-related acute toxicity, including laboratory abnormalities, must have recovered to CTCAE Grade 1 (v.4.0) or baseline, except toxicity not considered a safety risk.
* ECOG performance status of 0-2.
* Patient must have adequate organ function as determined by the following criteria:
* Serum creatinine ≤ 1.5 ULN or a calculated creatinine clearance of ≥ 50 mL/min
* Absolute neutrophil count ≥ 1.5 x 109/L
* Leukocytes > 3.0 x 109/L
* Hemoglobin > 80 g/L
* Platelets > 100 x 109/L
* Total bilirubin < ULN
* AST (SGOT) and ALT (SGPT) < 2.5 x ULN
* 12-Lead ECG with normal tracing, or clinically non-significant changes that do not require medical intervention
* QTc interval < 470 msec, and without history of Torsades de Pointes or other symptomatic QTc abnormality
* A normal LVEF of >50% as measured by ECHO or MUGA within 4 weeks prior to start of study treatment will be required for all patients

Exclusion Criteria:

* Patients who require segmental mandibulectomy for surgical resection of oral cavity tumor will not be enrolled
* Primary site of head and neck carcinoma in nasopharynx, skin, or unknown
* Prior or concurrent radiation therapy to tumor at site of planned resection
* Any clinically significant gastrointestinal abnormalities, which may impair intake, transit or absorption of PF-00299804
* Requirement for treatment with drugs that are highly dependent on CYP2D6 for metabolism since PF-00299804 is a potent CYP2D6 inhibitor in in vitro assays
* Patients currently taking drugs that have a risk of causing Torsades de Pointes
* Any acute or chronic medical, psychiatric condition or laboratory abnormality that could increase the risk associated with trial participation or trial drug administration or could interfere with interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry in the trial
* Other serious uncontrolled medical disorder or active infection that would impair the ability to receive study treatment as determined by investigator
* Dementia or significantly altered mental status that would limit the ability to obtain informed consent and compliance with the requirements of this protocol
* Patients breastfeeding or pregnant are excluded. All female patients with reproductive potential must have a negative pregnancy test within 72 hours prior to treatment.
* Patients of reproductive potential or their partners must agree to use effective contraception while receiving trial treatment and for at least 3 months thereafter.
* Current enrollment in another therapeutic clinical trial
* Inability/lack of willingness to comply with visits, treatment plans, protocol assessments or laboratory tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-05; Primary Completion 2012-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To assess the degree of modulation of the proliferation index, ki-67, in the primary tumor of OCC specimens following a short, preoperative course of PF-00299804 | 8-11 months

SECONDARY OUTCOMES:
To evaluate changes in tissue and blood-based biomarkers before, during and after treatment with PF-00299804 and attempt to correlate with gene expression changes, EGFR variant III mutation status, EGFR amplification and histopathological changes | 8-11 months
To assess the relationship between pharmacokinetic parameters and molecular changes detected in OCC tumor specimens | 8-11 months
To assess the safety and tolerability of pre-operative PF-00299804 | 8-11 months
To quantitatively assess the effect of PF-00299804 on tumorigenic cells expressing CD44+/Lin- markers in paired OCC tumor specimens | 8-11 months
To evaluate gene expression changes in tumor tissue before and after treatment with PF00299804 | 8-11 months

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, FRCPC, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada